CLINICAL TRIAL: NCT04106986
Title: The Effect Of Pulsed Electromagnetic Field And Progressive Resistance Exercise On Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43/120/2019
Record Dates: First submitted 2019-07-14; First posted 2019-09-27 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Pulsed Electromagnetic Field; Progressive Resistance Exercise
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized control trial study to investigate the effect of pulsed electromagnetic field and progressive resistance exercise on knee osteoarthritis regard pain level ,physical function, and quality of life
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and outcome assessor are blinded to subject assigned group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF and PRE (Experimental): The PEMF and PRE group received 24 sessions (3 sessions/week for 8 weeks) of combined treatment group (pulsed electromagnetic field with PRE training)
  Interventions: Combination Product: Pulsed electromagnetic field and Progressives resistance exercise
- PRE (Experimental): The PRE group received 24 sessions (3 sessions/week for 8 weeks) of only progressive resistance exercise
  Interventions: Other: PRE

INTERVENTIONS:
Combination Product: Pulsed electromagnetic field and Progressives resistance exercise — The pulsed electromagnetic field treatment consist of 30 minutes pulsed electromagnetic field with 50 Hz pulses
  The progressive resistance exercise training consist of 45 minutes of progressive resistance exercise protocol as the following:
  The PRE session begun with warm-up exercises that included riding a stationary ergometer for 5 minutes followed by stretching exercises for the hamstrings, quadriceps and gastrocnemius muscles. After this, subjects performed non-weight bearing (open chain) and weight bearing (closed chain) quadriceps exercises.
  The amount of resistance and number of repetitions for each exercise are based on a modification of the daily adjustable progressive resistance exercise (DAPRE) program that was described by Knight eta al.
  Arms: PEMF and PRE
Other: PRE — The progressive resistance exercise training consist of 45 minutes of progressive resistance exercise protocol as the following:
  The PRE session begun with warm-up exercises that included riding a stationary ergometer for 5 minutes followed by stretching exercises for the hamstrings, quadriceps and gastrocnemius muscles. After this, subjects performed non-weight bearing (open chain) and weight bearing (closed chain) quadriceps exercises.
  The amount of resistance and number of repetitions for each exercise are based on a modification of the daily adjustable progressive resistance exercise (DAPRE) program that was described by Knight eta al.
  Arms: PRE

SUMMARY:
The purpose of this study is to investigate the effect of pulsed electromagnetic field and progressive resistance exercise on Knee Osteoarthritis. It is experimental research study that look at the additive effect of pulsed electromagnetic field and progressive resistive exercise on pain level, patient-reported and performance-based physical function and Quality of life for patients with knee osteoarthritis

DETAILED DESCRIPTION:
Background: osteoarthritis is the main cause of disability in elderly population.[1,2] It affects almost one third of individuals aged 65 and older and approximately 25% of osteoarthritis patients 60 years and older cannot perform activities of daily living.[3] The clinical symptoms that lead to disability in Knee osteoarthritis are more frequent than all other joint complaint.

A large body of evidence exists proving the beneficial effects of progressive resistance exercise (PRE) in patients with knee osteoarthritis (OA).[4,5,6] Pulse electromagnetic field(PEMF) is a physical therapy modality that could be used for treating knee osteoarthritis (OA) and there emerging evidence suggesting its beneficial effect in reducing pain and improving function for knee osteoarthritis (OA)[7] The purpose of the study is to examine the effectiveness of using pulsed electromagnetic field (PEMF) with progressive resistance exercise (PRE) training in decreasing pain level ,improving physical function, and improving quality of life in patients with Knee osteoarthritis (OA) A small randomized control trial conducted to recruit 32 patients with knee osteoarthritis (OA). Participants with knee osteoarthritis (OA) as defined by American College of Rheumatology recruited from Prince Basma Educational Hospital. Eligible patients were randomly assigned to receive 24 sessions (3 sessions/week for 8 weeks) of either the combined (PRE and PEMF) treatment or PRE only. Participants will be evaluated at baseline, after the end of treatment protocol (8 weeks), and at 3 and 6 months follow up. Mixed ANOVA and repeated measure ANOVA will be used to evaluate the differences between groups in pain, and physical function, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* 40 year-old and above
* Diagnosed with unilateral or bilateral knee OA

Exclusion Criteria:

* Patients with current or previous knee surgeries
* Inflammatory arthritis's (rheumatoid arthritis, gout, etc.)
* Alzheimer disease
* Parkinson disease
* Unable to walk unaided for 6 months

To maximize the efficiency of our experiments we excluded patients if they:

* Have participated in progressive resistance training or received pulsed electromagnetic field treatment in the prior year
* Exercise regularly more than once a week.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Change Scores of The Knee Injury and Osteoarthritis Outcome Score | Baseline, 4 weeks, 3 and 6 month follow-up
  is knee-specific instrument , developed to assess the patients opinion about their knee and associated problems. the Knee Injury and osteoarthritis outcome Score(KOOS) evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored sub-scales; pain, other symptoms , functions in daily living (ADL), Function in sport and Recreation (sport/Rec), and knee-related Quality of Life (QOL). An Arabic version of KOOS has been found to be valid and reliable was used in our study[8]
Change Scores of The Short Physical Performance Battery (SPPB) | Baseline, 4 weeks, 3 and 6 month follow-up
  The SPPB assesses lower extremity function and has 3 components: walking gait speed, standing balance, and time to complete 5 chair stands. The total score is the sum of the three tests scores. The total score will be the variable used during data analysis. The SPPB has demonstrated good intra and inter-tester reliability, responsiveness, and validity[9,10]

SECONDARY OUTCOMES:
Change Scores of The Numeric pain rating scale (NPRS) | Baseline, 4 weeks, 3 and 6 month follow-up
  The NPRS is an 11-point scale comprising a number from 0 through 10; 0 indicates "no pain", and 10 indicates the "worst imaginable pain". Patients are instructed to choose a single number from the scale that best indicates their level of pain. The Arabic version of NPRS has shown good to excellent test-retest reliability and validity for patients with knee OA.[11]
Change Scores of The RAND-36 health survey | Baseline, 4 weeks, 3 and 6 month follow-up
  The RAND-36 (identical items of SF-36 health survey with different scoring system) is an easily administered health status and quality of life self-reported measure. It consists of 36-items that assess eight health concepts: general health perceptions, physical functioning, limitations of activities due to physical health problems, limitations of activities due to emotional problems, bodily pain, social functioning, energy and emotional well-being. A valid and reliable Arabic version of RAND-36 health survey was used in our study.[12]

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad, Irbid, Jordan

REFERENCES:
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Bijlsma JW, Berenbaum F, Lafeber FP. Osteoarthritis: an update with relevance for clinical practice. Lancet. 2011 Jun 18;377(9783):2115-26. doi: 10.1016/S0140-6736(11)60243-2. PMID 21684382
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Bartholdy C, Juhl C, Christensen R, Lund H, Zhang W, Henriksen M. The role of muscle strengthening in exercise therapy for knee osteoarthritis: A systematic review and meta-regression analysis of randomized trials. Semin Arthritis Rheum. 2017 Aug;47(1):9-21. doi: 10.1016/j.semarthrit.2017.03.007. Epub 2017 Mar 18. PMID 28438380
- [Background] Bennell KL, Dobson F, Hinman RS. Exercise in osteoarthritis: moving from prescription to adherence. Best Pract Res Clin Rheumatol. 2014 Feb;28(1):93-117. doi: 10.1016/j.berh.2014.01.009. PMID 24792947
- [Background] Loew L, Brosseau L, Kenny GP, Durand-Bush N, Poitras S, De Angelis G, Wells GA. An evidence-based walking program among older people with knee osteoarthritis: the PEP (participant exercise preference) pilot randomized controlled trial. Clin Rheumatol. 2017 Jul;36(7):1607-1616. doi: 10.1007/s10067-017-3606-9. Epub 2017 Mar 22. PMID 28332010
- [Background] Nicolakis P, Kollmitzer J, Crevenna R, Bittner C, Erdogmus CB, Nicolakis J. Pulsed magnetic field therapy for osteoarthritis of the knee--a double-blind sham-controlled trial. Wien Klin Wochenschr. 2002 Aug 30;114(15-16):678-84. PMID 12602111
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Alghadir AH, Anwer S, Iqbal ZA. The psychometric properties of an Arabic numeric pain rating scale for measuring osteoarthritis knee pain. Disabil Rehabil. 2016 Dec;38(24):2392-7. doi: 10.3109/09638288.2015.1129441. Epub 2016 Jan 6. PMID 26733318
- [Background] Coons SJ, Alabdulmohsin SA, Draugalis JR, Hays RD. Reliability of an Arabic version of the RAND-36 Health Survey and its equivalence to the US-English version. Med Care. 1998 Mar;36(3):428-32. doi: 10.1097/00005650-199803000-00018. PMID 9520966